CLINICAL TRIAL: NCT06615466
Title: Super-Hypofractionated Partial Breast Irradiation After Breast-Conserving Surgery for Early-Stage Low-Risk Breast Cancer: a Prospective, Single-arm Trial
Brief Title: Super-Hypofractionated Partial Breast Irradiation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-008224; 22/117-3318
Record Dates: First submitted 2024-04-18; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Partial Breast Irradiation (Experimental)
  Interventions: Radiation: Partial Breast Irradiation

INTERVENTIONS:
Radiation: Partial Breast Irradiation — 26Gy/5.2Gy/5f

SUMMARY:
Partial breast irradiation is currently a hot topic in clinical research, but the appropriate population and appropriate irradiation The technology and dose fractionation mode are still inconclusive. Foreign studies have mostly selected patients with low risk of recurrence. Breast-conserving surgeries for early-stage breast cancer are increasing year by year in China. It is necessary to conduct prospective clinical studies to explore the Chinese population suitable for partial breast irradiation and the appropriate radiotherapy dose fractionation model. A preliminary study in our center has compared the safety and efficacy of a 2-week schedule of partial breast irradiation (40Gy/10f) and a 3-week schedule of whole-breast radiotherapy (43.5Gy/15f) in patients with early-stage low-risk breast cancer after breast-conserving surgery. , preliminary results show that the 2-week partial breast irradiation regimen is safe and effective. This study plans to continue to select low-risk breast-conserving patients, use extracorporeal intensity-modulated radiotherapy technology, refer to the radiotherapy dose fractionation model of the FAST-Forward study, and give partial breast irradiation 5.2 Gy/f/d, a total of 5 times, with a total dose of 26Gy, to further shorten the time The radiotherapy time is 1 week, and the acute and late adverse reactions of radiotherapy and the local control of the tumor are prospectively observed. Provide evidence for conducting a national multi-center phase III clinical randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥45 years old, <75 years old women
2. Life expectancy >5 years
3. Start radiotherapy within 12 weeks after breast-conserving surgery (or within 8 weeks from the end of chemotherapy)
4. Invasive ductal carcinoma grade 1-2, or mucinous carcinoma, papillary carcinoma, canalicular carcinoma, medullary carcinoma; primary tumor

   ≤3.0cm; both pN0 (axillary dissection or sentinel lymph node biopsy)
5. Low-risk DCIS: tumor ≤2.5cm, low to medium grade; axillary surgery is not required or pN0
6. Single focus (with MRI diagnosis)
7. Vascular tumor thrombus negative
8. ER and/or PR positivity (defined as strong positivity in >1% of tumor cell nuclei)
9. Negative pathological margin≥2mm
10. Place metal markers on the tumor bed
11. Sign the informed consent form

Exclusion Criteria:

1. Multiple primary tumors
2. Invasive ductal carcinoma grade 3
3. Invasive micropapillary carcinoma
4. Lobular carcinoma in situ
5. Invasive lobular carcinoma
6. Simple nipple paget's disease
7. Oncoplastic surgery
8. Neoadjuvant chemotherapy or neoadjuvant endocrine therapy
9. Previous or simultaneous contralateral breast cancer
10. History of ipsilateral chest wall radiotherapy
11. Have active collagen vascular disease

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute adverse reactions | up to 6 months

SECONDARY OUTCOMES:
Incidence of late adverse reactions | through study completion, an average of 5 year
Survival | through study completion, an average of 5 year
  Local recurrence rate, regional recurrence rate, distant metastasis rate, disease-free survival rate and overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital ,National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided